CLINICAL TRIAL: NCT00005829
Title: Phase II Study of Gemcitabine for Relapsed B-Cell Chronic Lymphocytic Leukemia
Brief Title: Gemcitabine in Treating Patients With Recurrent Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-98-81-52; NCCTG-988152; CDR0000067843 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02331 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2000-06-02; First posted 2004-06-18 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 4 weeks for a minimum of 3 courses. Patients achieving clinical complete remission, complete remission, nodular partial remission, or partial remission following 3 courses of therapy, receive 2 additional courses of therapy. Patients achieving complete remission or further improvement following the 2 additional courses of therapy, receive another 2 courses of therapy. Patients are followed every 3 months until disease progression or relapse. Patients achieving complete remission are followed every 6 months for 1 year.
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine in treating patients who have recurrent chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rate and duration of complete and partial remission in patients with recurrent B-cell chronic lymphocytic leukemia treated with gemcitabine. II. Assess the toxicities of this regimen in these patients.

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 4 weeks for a minimum of 3 courses. Patients achieving clinical complete remission, complete remission, nodular partial remission, or partial remission following 3 courses of therapy, receive 2 additional courses of therapy. Patients achieving complete remission or further improvement following the 2 additional courses of therapy, receive another 2 courses of therapy. Patients are followed every 3 months until disease progression or relapse. Patients achieving complete remission are followed every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of B-cell chronic lymphocytic leukemia manifested by all of the following: Minimum threshold peripheral lymphocyte count of at least 5,000/mm3 Small to medium sized peripheral blood lymphocytes with no greater than 55% prolymphocytes Bone marrow aspirate and biopsy containing at least 30% lymphoid cells Immunophenotypic and biopsy evaluation of peripheral blood lymphocytes demonstrating monoclonality of B lymphocytes B-cell markers with CD5 antigen (e.g., T-1, T-101) in the absence of other pan T-cell markers (e.g., CD3, CD2) Expression of CD19, CD20, and CD23 B cell surface markers B-cell expression of kappa or lambda light chains Active disease with at least one of the following criteria: One or more disease related symptoms: At least 10% weight loss within the past 6 months Fever greater than 100.5 F for at least 2 weeks without evidence of infection Night sweats without evidence of infection Evidence of progressive marrow failure as manifested by the development of or worsening of anemia (hemoglobin less than 11.0 g/dL) and/or thrombocytopenia (platelet count less than 100,000/mm3) (i.e., any stage III or IV disease) Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroid therapy Massive (i.e., greater than 6 cm below the left costal margin) or progressive splenomegaly (i.e., a greater than 50% increase over two months) Massive (i.e., greater than 10 cm in longest diameter) or progressive lymphadenopathy (i.e., a greater than 50% increase over two months) Progressive lymphocytosis with an increase of greater than 50% over a 2 month period (unrelated to corticosteroids) or an anticipated doubling time of less than 6 months No marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any criteria for active disease Previously treated with at least a fludarabine or cladribine based regimen and a prior alkylating agent with evidence of recurrent or progressive disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Platelet count at least 75,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 1.5 times ULN (unless due to hemolysis or chronic lymphocytic leukemia) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease No myocardial infarction within the past month Other: No uncontrolled infection HIV negative No other active malignancy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy Endocrine therapy: See Disease Characteristics No concurrent corticosteroids Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2000-02; Primary Completion 2002-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
confirmed response | Up to 20 weeks

SECONDARY OUTCOMES:
overall survival | Up to 8 years
progression free survival | Up to 8 years
time to progression | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy G. Call, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Call TG, Constantinou CL, Kahanic SP, et al.: NCCTG trial of gemcitabine for relapsed B-cell chronic lymphocytic leukemia. [Abstract] J Clin Oncol 22 (Suppl 14): A-6726, 613s, 2004.